CLINICAL TRIAL: NCT02895516
Title: A Prospective, Open-label, Single-arm Study to Assess the Ease of Use, Tolerability, Efficacy and Safety of the Vibrant Capsule Administered in the Home Environment.
Brief Title: Ease of Use, Tolerability, Efficacy and Safety of the Vibrant Capsule Administered in the Home Environment
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Vibrant Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 230CLD
Record Dates: First submitted 2016-09-06; First posted 2016-09-09 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vibrating Capsule (Other): Patients will receive vibrating capsule for 6 weeks of treatment (2 capsules per week)
  Interventions: Device: Vibrating capsule

INTERVENTIONS:
Device: Vibrating capsule — Patients will receive vibrating capsule for 6 weeks of treatment (2 capsules per week)

SUMMARY:
The study is a prospective, open-label, single-arm study, to evaluate the ease of use, tolerability, efficacy and safety of the Vibrant Capsule administered in the home environment.

One arm will be assessed: Vibrant Capsule administered twice a week.

Patients will follow a 2 weeks baseline period and then take the Vibrant Capsule for a treatment period of 6 weeks.

During the 2 weeks of baseline, patients will be asked to refrain from taking any medication or supplement to relieve their constipation.

After 14 days the patients will return and eligibility will be re-assessed. Patients will be instructed to complete a simple patient eDiary each day throughout the duration of the study. After 3 weeks of treatment, the patient will attend for evaluation and to receive new capsules. A final visit will take place at the end of the 6 week treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 22 years and older
2. Patients with Chronic Idiopathic Constipation according to Rome III criteria and who have not experienced relief of their symptoms from available therapies (osmotic and stimulant laxatives used for at least one month at recommended dose)
3. Patients with an average of less than 3 Spontaneous Bowel Movements per week and at least 1 Spontaneous Bowel Movements per week
4. Normal colonoscopy performed within 10 years prior to study participation, unless the patients are less than 50 years old and without alarm signs and/or symptoms
5. Patient signed the Informed Consent Form
6. Female subjects must have a negative urine pregnancy test and must not be lactating prior to receiving study medication. For females of child-bearing potential, a hormonal (i.e., oral, implantable, or injectable) and single-barrier method, or a double-barrier method of birth control must be used throughout the study. All other female subjects must have the reason for their inability to bear children documented in the medical record [i.e., tubal ligation, hysterectomy, or post-menopausal (defined as a minimum of one year since the last menstrual period)]; in these circumstances, a urine pregnancy test will not be necessary.

Exclusion Criteria:

1. History of complicated/obstructive diverticular disease
2. History of intestinal or colonic obstruction, or suspected intestinal obstruction.
3. History of significant gastrointestinal disorder, including any form of inflammatory bowel disease or gastrointestinal malignancy (celiac disease is accepted if the subject has been treated and is in remission)
4. History of gastroparesis
5. Use of any of the following medications:

   * Medications that may affect intestinal motility, prokinetics, anti-depressants, anti-Parkinsonian medications, opiates, opioids, calcium-channel blockers, aluminum/magnesium hydroxide
   * With the exception of antidepressants, thyroid or hormonal replacement therapy, when the subject has been on a stable dose for at least 3 months prior to enrollment.
6. Clinical evidence of significant respiratory, cardiovascular, renal, hepatic, biliary, endocrine, psychiatric or neurologic disease.
7. Presence of cardiac pacemaker or gastric electrical stimulator.
8. History of, or current eating disorders, such as anorexia, bulimia, or compulsory overeating.
9. Diagnosis of mega-rectum or colon, congenital anorectal malformation, clinically significant rectocele, history of intestinal resection (with an exception for appendectomy, cholecystectomy and inguinal hernia repair), history of bariatric surgery or evidence of any structural abnormality of the gastrointestinal tract that might affect transit
10. History of Zenker's diverticulum, dysphagia, Barrett's esophagus, esophageal stricture or achalasia
11. Chronic use of non-steroidal anti-inflammatory drugs: chronic use is defined as taking full dose non-steroidal anti-inflammatory drugs more than three times a week for at least six months. Patients on cardiac doses of aspirin may be enrolled in the study
12. Patients with pelvic floor dysfunction/defecatory disorder, based on patient history
13. Participation in another clinical study within one month prior to screening.
14. Women who are pregnant or lactating
15. Use of any medication for constipation relief during the study, except as rescue medication, as indicated by study rules
16. Inability to use an electronic daily Diary (on a computer, phone application, tablet or other electronic device) to report bowel movements, symptoms and medication usage
17. Any other condition which in the opinion of the investigator may adversely affect the safety of the patient or would limit the patient's ability to complete the study

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10; Primary Completion 2017-04 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Spontaneous Bowel Movements success rate | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ashok Tuteja, MD, Principal Investigator — University of Utah Healthcare
Locations (1):
- University of Utah HealthCare, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No